CLINICAL TRIAL: NCT05891054
Title: Effects of the Inclusion of Physical Activity in Secondary School Academic Classes on Educational Indicators and Health Markers: the ACTIVE CLASS Study
Brief Title: Effects of the Inclusion of Physical Activity in Secondary School Academic Classes: the ACTIVE CLASS Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government); Regional Ministry of Economy, Knowledge, Enterprise and University of Andalucia (Unknown)
Responsible Party: Principal Investigator, David Sanchez Oliva, Assistant professor, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PID2019-104023RA-I00
Record Dates: First submitted 2023-05-11; First posted 2023-06-06 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2023-06

CONDITIONS: Physical Activity; Adolescents; Cognition; Physical Fitness
Keywords: Active break; Physically active learning; Academic indicators; Motivational variables; Sedentary time
MeSH Terms: conditions — Motor Activity; Sedentary Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active breaks (Experimental): Active breaks consist of short breaks during academic classes other than physical education that include moderate to vigorous physical activity, usually unrelated to curricular content.
  In this type of intervention, 2 active breaks are taken daily in a predetermined time slot. The development of each break is done through access to a specific digital platform where students follow the instructions of an avatar, which is in charge of guiding the realization of the active break. Each active rest involves a total of 4 minutes of activity, in which two sets of 20 seconds of work and 10 seconds of rest of four different exercises are performed, ending with a brief return to calm consisting of two deep breaths. The activities selected for each of the active breaks include aerobic and strengthening activities of moderate and vigorous intensity.
  Interventions: Behavioral: Active breaks
- Physically active learning (Experimental): Physically active learning consists of the incorporation of physical activity (usually of moderate-vigorous intensity) into the educational content taught in academic lessons that do not refer to physical education.
  This type of intervention is carried out once a week for 1 hour outside the classroom, where physical activity (through movement, jumping, strengthening exercises, throwing, etc.) is incorporated into academic mathematics classes.
  The mathematics teachers (with the support of the research team) are in charge of teaching the physically active classes. Prior to the development of each class, the research team, together with the mathematics teachers involved, meet and design the class according to the contents to be addressed.
  Interventions: Behavioral: Physically active learning
- Control Group (No Intervention): The control group will receive the usual academic classes without any methodological modification during the intervention period.

INTERVENTIONS:
Behavioral: Active breaks — Two active breaks are taken daily in a predetermined time slot. The development of each break is done through access to a specific digital platform where students follow the instructions of an avatar, which is in charge of guiding the realization of the active break. Each active rest involves a total of 4 minutes of activity, in which two sets of 20 seconds of work and 10 seconds of rest of four different exercises are performed, ending with a brief return to calm consisting of two deep breaths. The activities selected for each of the active breaks include aerobic and strengthening activities of moderate and vigorous intensity.
  Arms: Active breaks
Behavioral: Physically active learning — The physically active learning is carried out once a week for 1 hour outside the classroom, where physical activity (through movement, jumping, strengthening exercises, throwing, etc.) is incorporated into academic mathematics classes.
  The mathematics teachers (with the support of the research team) are in charge of teaching the physically active classes. Prior to the development of each class, the research team, together with the mathematics teachers involved, meet and design the class according to the contents to be addressed.
  Arms: Physically active learning

SUMMARY:
Study based on the inclusion of physical activity in the secondary education classroom through active breaks and physically active learning, aimed at testing its effects on the improvement of physical activity levels, sedentary time, educational indicators, cognition and physical and psychological health markers.

DETAILED DESCRIPTION:
The ACTIVE CLASS is a randomized controlled study coordinated by fully qualified researchers in the physical activity and sport sciences from two universities [University of Cadiz (UCA) and University of Extremadura (UEX), Spain]. This study is aimed at 7th and 8th grade students (11-13 years old), belonging to 6 schools in Spain (3 schools in Cadiz and 3 schools in Caceres). One school from each study region will be randomly assigned to one of the three intervention groups:

(i) Active breaks intervention: there will be 2 active breaks per day, 5 days a week of moderate-vigorous physical activity with a duration of 5 minutes.

(ii) Physically active learning intervention: Once a week, moderate-vigorous physical activity will be included in the academic lessons of the mathematics subject.

(iii) Control group.

The interventions will have a duration of 16 weeks. The different outcome measures (physical activity and sedentary behavior, health-related physical fitness, psychological health, academic indicators, cognition, motivational variables, dietary patterns, sociodemographic characteristics and qualitative information) will be evaluated at 3 time points:

1. Pre-intervention
2. Post-intervention
3. Retention measure (this measure will be conducted four weeks after the intervention to analyze the sustainability of the intervention program)

All measures will be assessed at each time point with the exception of qualitative information which will be assessed only in the post-intervention measure.

At the end of the intervention the researchers will determine the changes of the main outcome variables. Likewise, the main hypotheses raised will be:

1. A physically active learning intervention and active breaks will result in improved physical activity levels and decreased sedentary time.
2. A physically active learning intervention and active breaks will produce improvements in markers of physical and psychological health.
3. The inclusion of physical activity in academic classes will result in improved academic indicators and cognitive markers.
4. A physically active learning intervention and active breaks will produce improvements on motivational variables in academic classes.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents who are studying 7th or 8th grade
* Adolescents with the informed consent signed by family/tutor
* Schools with at least 60 students enrolled in 7th and/or 8th grade
* Schools belonging to the regions of Cáceres and Cádiz

Exclusion Criteria:

* Adolescents who have a physical disability or health condition that could limit physical activity levels
* Schools participating in any other physical activity or health promotion program

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 292 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Physical activity and sedentary time | 6 months
  Physical activity and sedentary time will be measured through accelerometry (Actigraph GT3X+, Inc., Pensacola, FL, USA).

SECONDARY OUTCOMES:
Cardiorespiratory capacity | 6 months
  The 20-metre shuttle run test will be used to assess cardiorespiratory fitness. Participants will run the 20-metre distance to the rhythm of a recording. The initial speed is 8.5 km/h and will be increased by 0.5 km/h per section. The race will end when the participant stops due to fatigue or when he/she fails to cross the marked lines to the rhythm of the acoustic signals on two consecutive occasions. The last stage or half stage completed by the competitor will be scored.
Musculoskeletal capacity of upper body | 6 months
  The hand grip test will be used to assess musculoskeletal capacity of upper body. The test shall be performed twice with each hand alternately. The maximum score of each hand in kilograms shall be recorded and the mean value between them shall be calculated.
Musculoskeletal capacity of lower body | 6 months
  Standing broad jump shall be used to assess the musculoskeletal capacity of the lower limbs. The participant shall stand behind a line with feet shoulder width apart. The participant is then asked to jump forward as far as possible with both feet. If he/she rests his/her hands or lifts his/her feet off the ground when landing, the test is invalid. The test shall be performed twice, and the best score recorded in centimetres.
Body mass index | 6 months
  Weight and height will be combined to report BMI in kg/m^2. In both cases the measurement shall be performed twice and the mean shall be recorded.
Body composition | 6 months
  Waist circumference shall be measured as a body composition variable with a non-elastic tape placed in the frontal plane at the midpoint between the upper iliac spine and the costal border at the mid-axillary line. The measurement shall be taken twice and the mean of the two measurements shall be recorded.
Subjective physical fitness | 6 months
  The International Fitness Scale will be used for the assessment of subjective physical fitness. Participants will be asked to rate each of the fitness components on a 5-point Likert-type scale ranging from: "very poor" (1); "poor" (2); "fair" (3); "good" (4) and "very good".
Health status | 6 months
  The EuroQol five dimensions three levels will be used to assessment of health status (EQ-5D-3L).This questionnaire is composed of the dimensions of: (i) mobility; (ii) self-care; (iii) usual activities; (iv) pain/discomfort and (v) anxiety/depression. The three levels that participants should mark a Likert-type scale correspond to (i) no problem; (ii) some problems; (iii) many problem.
Self-perceived health | 6 months
  Self-perceived health will be measured through the classic self-reported health item, where participants will have to classify their health among the following options: "excellent" (5); "very good" (4); "good" (3); "fair" (2) and "poor" (1).
School engagement | 6 months
  The engagement scale (UWES-S-9) will be used to evaluate school engagement. The UWES-S-9 is composed of nine items that reflect the three dimensions of engagement: (i) vigor; (ii) absorption; and (iii) dedication, each dimension is represented by three items that will be evaluated through a Likert-type scale, ranging from "never" (0 points) to "always" (6 points).
Learning perception | 6 months
  Learning perception in mathematics and in general studies will be assessed by means of a questionnaire consisting of eight items. Items 1- 4 will assess the "perceived learning" dimension and items 5-8 will measure the "satisfaction with learning" dimension. All items will be scored according to a five-point Likert scale, where "1" is (strongly disagree) and "5" is (strongly agree).
Academic performance | 6 months
  Academic performance will be evaluated through the marks reported by the schools before and after the intervention.
Time on task | 6 months
  Time on task will be assessed by direct observation in mathematics classes or in the classes were the active breaks take place, and in the consecutive class one hour later. Each researcher will assess a total of six students per assessment, where they have 15 seconds per subject to observe, identify the type of behaviour and record it on a worksheet. The researcher will repeat this process for the entire hour. Behaviours will be classified as 'on-task' and 'off-task'. The latter shall be divided into (i) "off-task-motor"; (ii) "off-task-noise"; (iii) "off-task-passive". The percentage of time students spend on each of the behaviours will be recorded.
Inhibition | 6 months
  Inhibition will be evaluated through the Flanker task protocol, part of the NIH Examiner programme. This is a computerised programme where the subject answers the tests individually. The algorithm provided by the program, ranging from 0 to 10, which includes accuracy and reaction time, will be recorded.
Cognitive flexibility | 6 months
  Cognitive flexibility will be evaluated through the Shifting task protocol, part of the NIH Examiner programme. This is a computerised programme where the subject answers the tests individually. The algorithm provided by the program, ranging from 0 to 10, which includes accuracy and reaction time, will be recorded.
Working memory | 6 months
  Working memory will be evaluated through the N-Back protocol, part of the NIH Examiner programme. This is a computerised programme where the subject answers the tests individually. The algorithm provided by the program, ranging from 0 to 10, which includes accuracy and reaction time, will be recorded.
Novelty | 6 months
  Novelty will be assessed through the Novelty Need Satisfaction Scale. Five of the 19 questions that make up the original scale will be selected and participants will be asked to answer them on a Likert-type scale where 1 = "strongly disagree" and 5 = "strongly agree".
Enjoyment and boredom | 6 months
  Enjoyment and boredom will be assessed using the Spanish version of The Sport Satisfaction Instrument. This scale is composed of eight items. Participants will have to rate their degree of agreement with the items referring to fun or boredom on a five-point Likert-type scale, ranging from 1 (strongly disagree) to 5 (strongly agree).
Dietary patterns | 6 months
  Adherence to the Mediterranean diet will be measured using the updated version 2.0 of the KIDMED questionnaire.
Sociodemographic characteristics | 6 months
  Sociodemographic characteristics will be measured through the Spanish-adapted version III of The Family Affluence Scale.
Teachers' and students' perception about the suitability and the development of physically active classes and active breaks | 6 months
  perception about the suitability and the development of physically active classes and active breaks (perceptions, barriers, points to improve, strengths...) a semi-structured interview will be conducted with the teachers involved in the intervention. Additionally, and for the same purpose, a discussion group will be developed for each of the proposed interventions with a subsample of students.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - University of Cádiz, Puerto Real, Cádiz
  - University of Extremadura, Cáceres

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grao-Cruces A, Martin-Acosta F, Vaquero-Solis M, Ruiz-Hermosa A, Camiletti-Moiron D, Sanchez-Oliva D. Fitness, Weight Status and Executive Functions in Adolescents: A Cluster Analysis. Scand J Med Sci Sports. 2025 Aug;35(8):e70098. doi: 10.1111/sms.70098. PMID 40719569
- [Derived] Gonzalez-Perez M, Sanchez-Oliva D, Grao-Cruces A, Cano-Canada E, Martin-Acosta F, Munoz-Gonzalez R, Bandera-Campos FJ, Ruiz-Hermosa A, Vaquero-Solis M, Padilla-Moledo C, Conde-Caveda J, Segura-Jimenez V, Gonzalez-Ponce I, Garcia-Calvo T, Castro-Pinero J, Camiletti-Moiron D. Effects of the inclusion of physical activity in secondary education academic classes on educational indicators and health markers: rationale and methods of the ACTIVE CLASS study. Front Public Health. 2024 Jan 5;11:1329245. doi: 10.3389/fpubh.2023.1329245. eCollection 2023. PMID 38249387